CLINICAL TRIAL: NCT04000568
Title: Breathing Pattern Variability in Preterm Infants: Effect of Non-invasive Neurally Adjusted Ventilatory Assist (NAVA-NIV) Versus Nasal Intermittent Positive Pressure Ventilation (PC-NIV), a Crossover Study
Brief Title: Breathing Variability and NAVA in Neonates
Acronym: BRAVe NANO
Status: Completed | Type: Observational
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Collaborators: Politecnico di Milano (Other)
Responsible Party: Principal Investigator, Anna Lavizzari, Principal Investigator, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Other Study IDs: BRAVe NANO (NIV)
Record Dates: First submitted 2019-05-31; First posted 2019-06-27 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Neonatal Respiratory Distress Syndrome; Prematurity
Keywords: Preterm Infant; Respiratory Distress Syndrome; Non-invasive respiratory Support; Neurally Adjust Respiratory Assist (NAVA); Nasal Intermittent Positive Pressure Ventilation
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn; Premature Birth; Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Population: All the infants enrolled in the study will receive 1 h of NAVA-NIV and 1h PC-NIV in a cross-over study design
  Interventions: Other: Respiratory support: NAVA -NIV and PC-NIV

INTERVENTIONS:
Other: Respiratory support: NAVA -NIV and PC-NIV — The infants enrolled will receive respiratory assistance by NAVA-NIV and PC-NIV in a randomized order

SUMMARY:
The current study is a crossover trial, aiming at evaluating the effect of NAVA -NIV compared to Nasal Intermittent Positive Pressure Ventilation (PC-NIV) at the same level of peak inspiratory pressure, in terms of: breath-by-breath variability of tidal breathing amplitude, variability of the other breathing patterns; lung mechanics; gas exchange; rate of episodes of apnea; bradycardia and desaturations; respiratory asynchrony and comfort, in preterm infants < 37+0 weeks+days post-menstrual age.

DETAILED DESCRIPTION:
Preterm infants matching the inclusion criteria (listed elsewhere) will be enrolled in a cross- over trial of two modes of non-invasive respiratory support: nasal intermittent positive pressure ventilation (PC-NIV) and NAVA NIV (Sevo-n Neonatal Ventilator, GETINGE, Solna, Sweden). Parental consent will be collected prior to the study. A 20-minute registration of ventilator parameters during assistance on NAVA-NIV will allow calculating the mean PIP (peak inspiratory pressure), in order to compare the two modes at the same level of PIP. The ventilator settings other than PIP (i.e. FiO2 (fraction of inspired oxygen), PEEP (positive end-expiratory pressure), IT (inspiratory time), RR (respiratory rate), NAVA level) will be based on the setting optimized by the attending physicians prior to the study entry. FiO2 will be adjusted in order to maintain SpO2 88-93% in infants ≤ 32 weeks of postconceptional age, 90-95% in infants > 32 weeks of postconceptional age. Infants will then receive a randomized sequence of 1-hour assistance by NAVA NIV and 1-hour assistance PC-NIV or vice-versa. Infants will receive respiratory support in a standardized supine position during the study period.

Two, high-resolution, small cameras will be placed in the infant's incubator to detect chest and abdominal movements, by means of two markers placed on the infant's chest and abdomen. Ventilators parameters (flow, pressure, volume, the electrical activity of the diaphragm), vital signs (SpO2, HR (heart rate), ABP( arterial blood pressure)), transcutaneous gases, changes in end-expiratory lung volume will be collected continuously. Episodes of apnea, bradycardia or desaturations and the number of interventions required by the nurses and the attending physicians during the study (e.g. adjustment of the interface, suctioning, interventions to provide comfort or optimize the respiratory support...) will be also collected during the study. Patients' comfort will be assessed at the end of each sequence by the attending nurse by means of the COMFORT scale. Lung mechanics will be measured at the end of each sequence by means of the Forced Oscillation Technique.

Data will be then analysed and compared offline.

ELIGIBILITY:
Inclusion Criteria:

* preterm birth < 37 weeks of gestational age
* need of non-invasive respiratory support
* parental consent

Exclusion Criteria:

* Major congenital abnormalities of the cardio-respiratory systems
* Severe Respiratory Failure requiring intubation and mechanical ventilation at the time of the study; pH < 7.25 pCO2> 65 mmHg; pulmonary hypertension of the newborn requiring pharmacological treatment (Nitric Oxide, Sildenafil)
* Hypoxic-Ischaemic Encephalopathy, neurological disorders which may compromise the integrity of the neural transmission from the brain to the diaphragm
* Contraindication to orogastric tube insertion (e.g. oesophageal atresia, gastric perforation...)
* Haemodynamic instability requiring inotropic agents
* Any condition that would expose the patient to undue risk as deemed by the attending physician

Ages: 1 Day to 3 Months | Sex: All
Age Groups: Child
Study Population: preterm infants born < 37 weeks of gestation, requiring non-invasive respiratory support
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2019-05-02 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Change in breath-by-breath variability of tidal breathing amplitude | over the last 30 minutes of each step (crossover trial, 2 steps, 1 hour-step)
  Tidal breathing amplitude will be recorded continuously by mean of two, high-resolution cameras placed inside the infant's incubator and skin (non-invasive) markers. Data will be analysed a posteriori applying the DFA (Detrended Fluctuation Analysis) technique.

SECONDARY OUTCOMES:
Respiratory Rate | at the beginning of the study, at 10minutes, 20minutes, 30minutes, 35minutes, 40minutes, 45minutes, 50minutes, 55minutes, for each step, in a 2-step crossover trial, 1-hour step
  Respiratory rate (breaths/min) will be recorded from the ventilator
Inspiratory Time | at the beginning of the study, at 10minutes, 20minutes, 30minutes, 35minutes, 40minutes, 45minutes, 50minutes, 55minutes, for each step, in a 2-step crossover trial, 1-hour step
  Inspiratory time (msec) will be recorded from the ventilator tracing
Duty Cycle | at the beginning of the study, at 10minutes, 20minutes, 30minutes, 35minutes, 40minutes, 45minutes, 50minutes, 55minutes, for each step, in a 2-step crossover trial, 1-hour step
  Duty Cycle (Inspiratory Time/ Total Time), will be calculated from the ventilator tracing
Total Respiratory System Oscillatory Resistance | at the end of each 1-hour step of the trial (crossover trial, 2 steps, 1 hour-step)
  Total Respiratory System Oscillatory Resistance will be measured by the Forced Oscillation Technique (FOT) at the end of each step, by superimposing to the ventilator waveform an oscillatory pressure of small amplitude at 10 Hz (Fabian, ACUTRONIC Medical Systems AG, Switzerland).
Total Respiratory System Oscillatory Reactance | at the end of each 1-hour step of the trial (crossover trial, 2 steps, 1 hour-step)
  Total Respiratory System Oscillatory Reactance will be measured by the Forced Oscillation Technique (FOT) at the end of each step, by superimposing to the ventilator waveform an oscillatory pressure of small amplitude at 10 Hz (Fabian, ACUTRONIC Medical Systems AG, Switzerland).
SpO2/FiO2 (Fraction on inspired oxygen) | at the beginning of the study, at 10minutes, 20minutes, 30minutes, 35minutes, 40minutes, 45minutes, 50minutes, 55minutes, for each step, in a 2-step crossover trial, 1-hour step
  SpO2 and FiO2 will be monitored continuously and FiO2 will be adjusted to the target SpO2 88-93% in infants ≤ 32 weeks of postconceptional age, SpO2 90-95% in infants > 32 weeks of postconceptional age.
tpCO2, Transcutaneous Carbon Dioxide Partial Pressure (mmHg) | at the beginning of the study, at 10minutes, 20minutes, 30minutes, 35minutes, 40minutes, 45minutes, 50minutes, 55minutes, for each step, in a 2-step crossover trial, 1-hour step
  tpCO2 will be monitrored continuously over the study period and recorded at specific time points
Rate of apneas, desaturations, bradycardias | over 1 hour, for each step (in a 2-step crossover trial, 1-hour step)
  Episodes of apnoeas, desaturations, bradycardias will be recorded over each study period
Rate of patient-ventilator asynchronies | over 1 hour, for each step (in a 2-step crossover trial, 1-hour step)
  Patient-ventilator asynchronies will be calculated by continuous recording of ventilator parameters (flow, pressure, volume and electrical diaphragmatic activity) and by continuous recording of abdominal and chest movements by high resolution cameras placed in the incubators and skin markers on abdomen and chest

OTHER OUTCOMES:
Patient's comfort: COMFORT-B scale | at the end of each 1-hour step
  Patient's comfort will be assessed by the attending nurse at the end of each step by means of the COMFORT-B scale (COMFORT behavioural scale). The COMFORT-B scale is a validated tool for assessing patients' comfort in Pediatric Intensive Care Unit.It includes the following items for comfort evaluation: alertness, calmness, respiratory response, cry, physical movements, muscle tone, facial tension. For each item a descriptive scale form 1 (the best) to 5 (the worst) is indicated and the operator can choose what is the most appropriate for the patient.
Number of caregivers interventions required | at the end of each 1-hour step
  The number of interventions required to the attending personnel during each step will be also recorded: for instance interventions to improve comfort, to adjust the ventilator interface, to optimize the efficacy of respiratory support, suctioning ...

CONTACTS AND LOCATIONS:
Overall Officials: Anna Lavizzari, MD, Principal Investigator — Fondazione IRCCS Cà Granda, Ospedale Maggiore Policlinico
Locations (1):
- NICU, Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: Yes
the study protocol, statistical analysis plan an Informed Consent (only in the original language, available in English under request) will be available from the study protocol submission date. Analytic code status: still undecided.
Supporting Information: Study Protocol, SAP
Time Frame: at protocol submission
Access Criteria: free

REFERENCES:
- [Background] Costeloe K, Hennessy E, Gibson AT, Marlow N, Wilkinson AR. The EPICure study: outcomes to discharge from hospital for infants born at the threshold of viability. Pediatrics. 2000 Oct;106(4):659-71. doi: 10.1542/peds.106.4.659. PMID 11015506
- [Background] Ancel PY, Goffinet F; EPIPAGE-2 Writing Group; Kuhn P, Langer B, Matis J, Hernandorena X, Chabanier P, Joly-Pedespan L, Lecomte B, Vendittelli F, Dreyfus M, Guillois B, Burguet A, Sagot P, Sizun J, Beuchee A, Rouget F, Favreau A, Saliba E, Bednarek N, Morville P, Thiriez G, Marpeau L, Marret S, Kayem G, Durrmeyer X, Granier M, Baud O, Jarreau PH, Mitanchez D, Boileau P, Boulot P, Cambonie G, Daude H, Bedu A, Mons F, Fresson J, Vieux R, Alberge C, Arnaud C, Vayssiere C, Truffert P, Pierrat V, Subtil D, D'Ercole C, Gire C, Simeoni U, Bongain A, Sentilhes L, Roze JC, Gondry J, Leke A, Deiber M, Claris O, Picaud JC, Ego A, Debillon T, Poulichet A, Coline E, Favre A, Flechelles O, Samperiz S, Ramful D, Branger B, Benhammou V, Foix-L'Helias L, Marchand-Martin L, Kaminski M. Survival and morbidity of preterm children born at 22 through 34 weeks' gestation in France in 2011: results of the EPIPAGE-2 cohort study. JAMA Pediatr. 2015 Mar;169(3):230-8. doi: 10.1001/jamapediatrics.2014.3351. PMID 25621457
- [Background] Hennessy EM, Bracewell MA, Wood N, Wolke D, Costeloe K, Gibson A, Marlow N; EPICure Study Group. Respiratory health in pre-school and school age children following extremely preterm birth. Arch Dis Child. 2008 Dec;93(12):1037-43. doi: 10.1136/adc.2008.140830. Epub 2008 Jun 18. PMID 18562451
- [Background] Doyle LW, Carse E, Adams AM, Ranganathan S, Opie G, Cheong JLY; Victorian Infant Collaborative Study Group. Ventilation in Extremely Preterm Infants and Respiratory Function at 8 Years. N Engl J Med. 2017 Jul 27;377(4):329-337. doi: 10.1056/NEJMoa1700827. PMID 28745986
- [Background] Dumpa V, Bhandari V. Surfactant, steroids and non-invasive ventilation in the prevention of BPD. Semin Perinatol. 2018 Nov;42(7):444-452. doi: 10.1053/j.semperi.2018.09.006. Epub 2018 Oct 2. PMID 30343941
- [Background] Bhandari V. The potential of non-invasive ventilation to decrease BPD. Semin Perinatol. 2013 Apr;37(2):108-14. doi: 10.1053/j.semperi.2013.01.007. PMID 23582965
- [Background] Morley CJ, Davis PG, Doyle LW, Brion LP, Hascoet JM, Carlin JB; COIN Trial Investigators. Nasal CPAP or intubation at birth for very preterm infants. N Engl J Med. 2008 Feb 14;358(7):700-8. doi: 10.1056/NEJMoa072788. PMID 18272893
- [Background] SUPPORT Study Group of the Eunice Kennedy Shriver NICHD Neonatal Research Network; Finer NN, Carlo WA, Walsh MC, Rich W, Gantz MG, Laptook AR, Yoder BA, Faix RG, Das A, Poole WK, Donovan EF, Newman NS, Ambalavanan N, Frantz ID 3rd, Buchter S, Sanchez PJ, Kennedy KA, Laroia N, Poindexter BB, Cotten CM, Van Meurs KP, Duara S, Narendran V, Sood BG, O'Shea TM, Bell EF, Bhandari V, Watterberg KL, Higgins RD. Early CPAP versus surfactant in extremely preterm infants. N Engl J Med. 2010 May 27;362(21):1970-9. doi: 10.1056/NEJMoa0911783. Epub 2010 May 16. PMID 20472939
- [Background] Arold SP, Suki B, Alencar AM, Lutchen KR, Ingenito EP. Variable ventilation induces endogenous surfactant release in normal guinea pigs. Am J Physiol Lung Cell Mol Physiol. 2003 Aug;285(2):L370-5. doi: 10.1152/ajplung.00036.2003. PMID 12851212
- [Background] Arold SP, Mora R, Lutchen KR, Ingenito EP, Suki B. Variable tidal volume ventilation improves lung mechanics and gas exchange in a rodent model of acute lung injury. Am J Respir Crit Care Med. 2002 Feb 1;165(3):366-71. doi: 10.1164/ajrccm.165.3.2010155. PMID 11818322
- [Background] Bellardine CL, Hoffman AM, Tsai L, Ingenito EP, Arold SP, Lutchen KR, Suki B. Comparison of variable and conventional ventilation in a sheep saline lavage lung injury model. Crit Care Med. 2006 Feb;34(2):439-45. doi: 10.1097/01.ccm.0000196208.01682.87. PMID 16424726
- [Background] Thammanomai A, Hueser LE, Majumdar A, Bartolak-Suki E, Suki B. Design of a new variable-ventilation method optimized for lung recruitment in mice. J Appl Physiol (1985). 2008 May;104(5):1329-40. doi: 10.1152/japplphysiol.01002.2007. Epub 2008 Mar 13. PMID 18339891
- [Background] Berry CA, Suki B, Polglase GR, Pillow JJ. Variable ventilation enhances ventilation without exacerbating injury in preterm lambs with respiratory distress syndrome. Pediatr Res. 2012 Oct;72(4):384-92. doi: 10.1038/pr.2012.97. Epub 2012 Jul 17. PMID 22805999
- [Background] Bartolak-Suki E, Noble PB, Bou Jawde S, Pillow JJ, Suki B. Optimization of Variable Ventilation for Physiology, Immune Response and Surfactant Enhancement in Preterm Lambs. Front Physiol. 2017 Jun 23;8:425. doi: 10.3389/fphys.2017.00425. eCollection 2017. PMID 28690548
- [Background] Arold SP, Malavia N, George SC. Mechanical compression attenuates normal human bronchial epithelial wound healing. Respir Res. 2009 Feb 12;10(1):9. doi: 10.1186/1465-9921-10-5. PMID 19171062
- [Background] Arold SP, Bartolak-Suki E, Suki B. Variable stretch pattern enhances surfactant secretion in alveolar type II cells in culture. Am J Physiol Lung Cell Mol Physiol. 2009 Apr;296(4):L574-81. doi: 10.1152/ajplung.90454.2008. Epub 2009 Jan 9. PMID 19136581
- [Background] Stein H, Firestone K. Application of neurally adjusted ventilatory assist in neonates. Semin Fetal Neonatal Med. 2014 Feb;19(1):60-9. doi: 10.1016/j.siny.2013.09.005. Epub 2013 Nov 13. PMID 24238745
- [Background] Stein H, Beck J, Dunn M. Non-invasive ventilation with neurally adjusted ventilatory assist in newborns. Semin Fetal Neonatal Med. 2016 Jun;21(3):154-61. doi: 10.1016/j.siny.2016.01.006. Epub 2016 Feb 16. PMID 26899957
- [Background] Firestone KS, Beck J, Stein H. Neurally Adjusted Ventilatory Assist for Noninvasive Support in Neonates. Clin Perinatol. 2016 Dec;43(4):707-724. doi: 10.1016/j.clp.2016.07.007. PMID 27837754
- [Background] Stein H, Alosh H, Ethington P, White DB. Prospective crossover comparison between NAVA and pressure control ventilation in premature neonates less than 1500 grams. J Perinatol. 2013 Jun;33(6):452-6. doi: 10.1038/jp.2012.136. Epub 2012 Oct 25. PMID 23100042
- [Background] Longhini F, Ferrero F, De Luca D, Cosi G, Alemani M, Colombo D, Cammarota G, Berni P, Conti G, Bona G, Della Corte F, Navalesi P. Neurally adjusted ventilatory assist in preterm neonates with acute respiratory failure. Neonatology. 2015;107(1):60-7. doi: 10.1159/000367886. Epub 2014 Nov 7. PMID 25401284
- [Background] de la Oliva P, Schuffelmann C, Gomez-Zamora A, Villar J, Kacmarek RM. Asynchrony, neural drive, ventilatory variability and COMFORT: NAVA versus pressure support in pediatric patients. A non-randomized cross-over trial. Intensive Care Med. 2012 May;38(5):838-46. doi: 10.1007/s00134-012-2535-y. Epub 2012 Apr 6. PMID 22481227
- [Background] Gibu CK, Cheng PY, Ward RJ, Castro B, Heldt GP. Feasibility and physiological effects of noninvasive neurally adjusted ventilatory assist in preterm infants. Pediatr Res. 2017 Oct;82(4):650-657. doi: 10.1038/pr.2017.100. Epub 2017 Jul 12. PMID 28399118
- [Background] Lee J, Kim HS, Jung YH, Shin SH, Choi CW, Kim EK, Kim BI, Choi JH. Non-invasive neurally adjusted ventilatory assist in preterm infants: a randomised phase II crossover trial. Arch Dis Child Fetal Neonatal Ed. 2015 Nov;100(6):F507-13. doi: 10.1136/archdischild-2014-308057. Epub 2015 Jul 15. PMID 26178463
- [Background] Baudin F, Wu HT, Bordessoule A, Beck J, Jouvet P, Frasch MG, Emeriaud G. Impact of ventilatory modes on the breathing variability in mechanically ventilated infants. Front Pediatr. 2014 Nov 25;2:132. doi: 10.3389/fped.2014.00132. eCollection 2014. PMID 25505779
- [Background] Garcia-Munoz Rodrigo F, Urquia Marti L, Galan Henriquez G, Rivero Rodriguez S, Hernandez Gomez A. Neural breathing patterns in preterm newborns supported with non-invasive neurally adjusted ventilatory assist. J Perinatol. 2018 Sep;38(9):1235-1241. doi: 10.1038/s41372-018-0152-5. Epub 2018 Jun 18. PMID 29910465
- [Background] Zannin E, Veneroni C, Dellaca RL, Corbetta R, Suki B, Tagliabue PE, Ventura ML. Effect of continuous positive airway pressure on breathing variability in early preterm lung disease. Pediatr Pulmonol. 2018 Jun;53(6):755-761. doi: 10.1002/ppul.24017. Epub 2018 Apr 23. PMID 29687665
- [Background] Peng CK, Havlin S, Stanley HE, Goldberger AL. Quantification of scaling exponents and crossover phenomena in nonstationary heartbeat time series. Chaos. 1995;5(1):82-7. doi: 10.1063/1.166141. PMID 11538314

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-27): https://cdn.clinicaltrials.gov/large-docs/68/NCT04000568/Prot_SAP_000.pdf